CLINICAL TRIAL: NCT07241845
Title: Epiretinal Membrane in Patients With Diabetic Retinopathy.
Brief Title: Epiretinal Membrane in Patients With DR.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Merna Maged Monir Aziz, resident doctor, Assiut University
Other Study IDs: epiretinal membrane in OCT
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Epiretinal Membrane
Keywords: oct
MeSH Terms: conditions — Epiretinal Membrane; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: OCT — All the patients will undergo OCT imaging using NIDEK RS-330 Retina scan duo 2 (SD-OCT)(CO-LTD made in Japan 2017) with scan speed 70.000 axial scans per second and wavelength of 880 nm. A three-dimensional scan protocol will be used for macular measurements. Macular scans will be performed with axial scanning protocols covering a 9 × 9 mm area centered on the fovea.
  OCT images will be evaluated by a trained ophthalmologist for the following:
  - Stage of ERM will be classified by Govetto et al system into stage 1,2,3 or 4.
  Stage 1: ERMs were mild and thin. Foveal depression is present. Stage 2: ERMs with a widening of the outer nuclear layer and loss of the foveal depression.
  Stage 3: ERMs with continuous ectopic inner foveal layers crossing the entire foveal area.
  Stage 4: ERMs were thick with continuous ectopic inner foveal layers and disrupted retinal layers.
  - central macular thickness CMT

SUMMARY:
To report the prevalence of ERM among patients with diabetic retinopathy, and the possible associated risk factors.

DETAILED DESCRIPTION:
Epiretinal membrane (ERM) can be defined as pre-retinal proliferation of myofibroblastic cells associated with extracellular matrix (ECM). Various aetiologies can lead to this final common pathway. Current imaging modalities are excellent at identifying and grading severity of ERMs, but do not yet differentiate histopathological variations which suggest that this is a heterogeneous group of diseases.

The prevalence of epiretinal membrane (ERM) is 7% to 11.8%, with increasing age being the most important risk factor. Although most ERM is idiopathic, common secondary causes include cataract surgery, retinal vascular disease, uveitis and retinal tears. Anti-VEGF injections are identified as a significant risk factor for ERM formation especially in patients with diabetes. The myofibroblastic pre-retinal cells are thought to transdifferentiate from glial and retinal pigment epithelial cells that reach the retinal surface via defects in the internal limiting membrane (ILM) or from the vitreous cavity. Grading schemes have evolved from clinical signs to ocular coherence tomography (OCT) based classification with associated features such as the cotton ball sign. Features predictive of better prognosis include absence of ectopic inner foveal layers, cystoid macular oedema, acquired vitelliform lesions and ellipsoid and cone outer segment termination defects. OCT-angiography shows reduced size of the foveal avascular zone.

The presence of continuous ectopic inner foveal layers was significantly associated with lower visual acuity. ERMs are divided into 4 stages. Stage 1 ERMs are mild and thin and a foveal depression was present. Stage 2 ERMs are associated with widening of the outer nuclear layer and loss of the foveal depression.

Stage 3 ERMs are associated with continuous ectopic inner foveal layers crossing the entire foveal area. In stages 1, 2, and 3 all retinal layers were clearly defined on OCT. Stage 4 ERMs are thick and associated with continuous ectopic inner foveal layers. In addition, retinal layers were disrupted.

Vitrectomy with membrane peeling remains the mainstay of treatment for symptomatic ERMs. Additional ILM peeling reduces recurrence but is associated with anatomical changes including inner retinal dimpling.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Patients with ERM confirmed by OCT images.
* Patients with DM with varying severity of diabetic retinopathy.

Exclusion Criteria:

* • History of previous eye trauma or surgery other than uneventful cataract surgery, uveitis, history of retinal detachment, media opacity impairing the quality OCT images, high myopia, macular or retinal diseases disease affecting the visual acuity other than diabetic retinopathy, e.g. macular hole, retinitis pigmentosa, AMD, CRVO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: diabetic patients above 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
frequency of ERM among patients presented with diabetic retinopathy | one year

SECONDARY OUTCOMES:
detection of possible associated risk factors including age, gender, type and duration and control of diabetes, hypertension, IHD, diabetic nephropathy, severity of diabetic retinopathy. | two years

REFERENCES:
- [Background] Kakihara S, AbdelSalam M, Zhuang K, Fawzi AA. Epiretinal Membrane Is Associated with Diabetic Retinopathy Severity and Cumulative Anti-VEGF Injections. Ophthalmol Sci. 2025 Feb 7;5(3):100733. doi: 10.1016/j.xops.2025.100733. eCollection 2025 May-Jun. PMID 40161463
- [Background] Bu SC, Kuijer R, Li XR, Hooymans JM, Los LI. Idiopathic epiretinal membrane. Retina. 2014 Dec;34(12):2317-35. doi: 10.1097/IAE.0000000000000349. PMID 25360790